CLINICAL TRIAL: NCT02479243
Title: Arterial Spin Labeling MRI Assessment and Quantification of Collateral Circulation in Unilateral Middle Cerebral Artery Atherosclerotic Stenosis
Brief Title: Assessment and Quantification of Collateral by ASL MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Deputy Chief of Radiology Department, Chinese PLA General Hospital
Other Study IDs: Xin Lou-ChinaPLAGH; Jh Lyu (Other: Chinese PLA General Hospital)
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Stroke
Keywords: Arterial Spin Labeling; MRI; Atherosclerotic Stenosis; Collateral Circulation; Ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Collateral Circulation: Symptomatic patients with unilateral MCA severe stenosis confirmed ≥ 90% by magnetic resonance angiography or 70-99% by conventional angiography were performed 3D pseudo-Continuous Arterial Spin Labeling MRI.

SUMMARY:
Collateral circulation supports brain tissues to maintain blood perfusion in cerebral ischemic stroke and are of great benefit for a better outcome. A non-invasive approach relative to currently widely used digital subtraction angiography (DSA) is needed. ASL (arterial spin labeling) is a novel perfusion method without contrast agent injection and features both temporal and cerebral blood flow(CBF) information. The investigators applied multiple post labeled delay(PLD) time to pseudo-continuous Arterial Spin Labeling (3D pCASL) MRI and subtraction images were obtained to evaluate the collateral robustness and quantitatively assess the collateral perfusion in patients with unilateral middle cerebral artery atherosclerotic stenosis and the ability to predict future stroke recurrence.

DETAILED DESCRIPTION:
Patients with unilateral middle cerebral artery (MCA) moderate to severe stenosis were consecutively enrolled. MRI protocols including diffusion weighted image, magnetic resonance angiography , 3D pCASL with two PLD of 1.5s and 2.5s were performed.

Cerebral blood flow(CBF) map of 3D pCASL with PLD 1.5s and 2.5s were postprocessed on workstation. Subtraction images were obtained by CBF 2.5s subtracted CBF 1.5s. Slices involving MCA downstream territory were equally separated as upper slices,middle slices and inferior slices corresponding to CIS system referring to previous study of Al-Ali F. Slices with residual signal areas more than 1/3 MCA territory involved would count 1, or would be 0. Total ASL collateral score(ASLCS) was calculated from 0-3. Then ,favorable collaterals were graded as total ASLCS 2-3 and poor collaterals were graded as total ASLCS 0-1.

Early-arriving flow perfusion proportion was defined as [CBF 1.5s at lesion side/CBF 2.5s of the contralateral side]×100%. Late-arriving perfusion proportion was defined as [(CBF 2.5s minus CBF 1.5s) at lesion side minus (CBF 2.5s minus CBF 1.5s) at normal side]/CBF 2.5s at the contralateral side ×100%. Antegrade scales and collateral grades were evaluated in patients with conventional angiography. Spearman correlation was analyzed between early-arriving and late-arriving flow and angiographic antegrade and collateral scales.

Baseline characteristics of patients were recorded including age, gender, hypertension,hypercholesterolemia,diabetes mellitus,smoking,obesity,qualifying stroke event, admission National Institute of Health stroke scale (NIHSS), diffusion-weighted image-ASPECTS.

One year stroke event recurrence and three months modified Rankin Scale (mRS) were followed up by neurologist by phone call or face to face.

Multi-variants Logistic Regression is performed to exam whether ASL collateral score and collateral perfusion quantification is significantly correlated with future ischemic event and functional outcome.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke or TIA in anterior circulation within 90 days
* MCA atherosclerotic moderate to severe stenosis(50%-99%) confirmed by conventional angiography or magnetic resonance angiography
* Age >18
* 2 or more atherosclerotic risk factors including hypertension, hypercholesterolemia, diabetes mellitus, cigarette smoking, and obesity
* Medical treatment
* Not receiving stent therapy
* Ability to comply with all studies

Exclusion Criteria:

* Multiple intracranial arteries stenosis (> 50%) or occlusion
* Less than 2 atherosclerotic risk factors
* Pregnancy and other contraindication to MRI scan
* Informed consent not obtained

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic and asymptomatic patients with MCA atherosclerotic moderate to severe stenosis(500%-99%) confirmed by conventional angiography or magnetic resonance angiography.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Stroke Event | Up to 1 year
  The patients were monitored whether they recured ischemic stroke event including transient ischemic attack (TIA) or stroke confirmed by neurologist and diffusion-weighted image MRI.

SECONDARY OUTCOMES:
modified Rankin Score | 3 months
  mRS of patients with acute or subacute stroke after 3 months were followed up for neurological outcome assessment. mRS < 2 was defined as favorable neurological outcome and mRS ≥ 2 was defined as poor neurological outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, MD, PHD., Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zaidat OO, Yoo AJ, Khatri P, Tomsick TA, von Kummer R, Saver JL, Marks MP, Prabhakaran S, Kallmes DF, Fitzsimmons BF, Mocco J, Wardlaw JM, Barnwell SL, Jovin TG, Linfante I, Siddiqui AH, Alexander MJ, Hirsch JA, Wintermark M, Albers G, Woo HH, Heck DV, Lev M, Aviv R, Hacke W, Warach S, Broderick J, Derdeyn CP, Furlan A, Nogueira RG, Yavagal DR, Goyal M, Demchuk AM, Bendszus M, Liebeskind DS; Cerebral Angiographic Revascularization Grading (CARG) Collaborators; STIR Revascularization working group; STIR Thrombolysis in Cerebral Infarction (TICI) Task Force. Recommendations on angiographic revascularization grading standards for acute ischemic stroke: a consensus statement. Stroke. 2013 Sep;44(9):2650-63. doi: 10.1161/STROKEAHA.113.001972. Epub 2013 Aug 6. No abstract available. PMID 23920012
- [Background] Al-Ali F, Jefferson A, Barrow T, Cree T, Louis S, Luke K, Major K, Nemeth D, Smoker S, Walker S. The capillary index score: rethinking the acute ischemic stroke treatment algorithm. Results from the Borgess Medical Center Acute Ischemic Stroke Registry. J Neurointerv Surg. 2013 Mar;5(2):139-43. doi: 10.1136/neurintsurg-2011-010146. Epub 2012 Jan 19. PMID 22266703
- [Background] Liebeskind DS, Cotsonis GA, Saver JL, Lynn MJ, Cloft HJ, Chimowitz MI; Warfarin-Aspirin Symptomatic Intracranial Disease (WASID) Investigators. Collateral circulation in symptomatic intracranial atherosclerosis. J Cereb Blood Flow Metab. 2011 May;31(5):1293-301. doi: 10.1038/jcbfm.2010.224. Epub 2010 Dec 15. PMID 21157476
- [Background] Liebeskind DS, Cotsonis GA, Saver JL, Lynn MJ, Turan TN, Cloft HJ, Chimowitz MI; Warfarin-Aspirin Symptomatic Intracranial Disease (WASID) Investigators. Collaterals dramatically alter stroke risk in intracranial atherosclerosis. Ann Neurol. 2011 Jun;69(6):963-74. doi: 10.1002/ana.22354. Epub 2011 Mar 17. PMID 21437932
- [Derived] Lyu J, Ma N, Liebeskind DS, Wang DJ, Ma L, Xu Y, Wang T, Miao Z, Lou X. Arterial Spin Labeling Magnetic Resonance Imaging Estimation of Antegrade and Collateral Flow in Unilateral Middle Cerebral Artery Stenosis. Stroke. 2016 Feb;47(2):428-33. doi: 10.1161/STROKEAHA.115.011057. Epub 2016 Jan 5. PMID 26732570